CLINICAL TRIAL: NCT00756886
Title: Does Atorvastatin Prevent Post Operative Atrial Fibrillation After Pulmonary Resection: A Randomized Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: F080722005
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2012-12

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Active Comparator): 40 mg QD for 7 days prior to surgery, and then continue at same dosage for 14 days after surgery.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): 40 mg QD for 7 days prior to surgery, and then continue at same dosage for 14 days after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 40 mg QD 7 day continue after procedure for 14 days
  Arms: Atorvastatin
Drug: Placebo — 40 mg QD for 7 days prior to surgery, and then continue at same dosage for 14 days after surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if atorvastatin (Lipitor) reduces the occurence of abnormal heart rhythm (atrial arrhythmia) following non cardiac thoracic surgery.

DETAILED DESCRIPTION:
The incidence of atrial arrhythmia after thoracic, non-cardiac procedures is exceedingly common and has been reported to occur in between 10-39% of patients. It has been shown to increase majority morbidity and also delay hospital discharge. Recent studies suggest that one week of pre-operative atorvastatin may reduce the incidence of post-operative atrial arrhythmia in patients who undergo cardiac surgery and a multi-institutional study is currently underway to further examine this concept. However, there are no published prospective randomized studies to date that have evaluated the effectiveness of atorvastatin to reduce atrial arrhythmia in patients who undergo thoracic, non-cardiac operations such as esophagectomy or pulmonary resection. The object of this study is to determine if atorvastatin reduces the incidence of atrial arrhythmia (atrial fibrillation or flutter) following non-cardiac thoracic surgery, specifically pulmonary resections.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective non-cardiac thoracic surgery requiring thoracotomy for resection

Exclusion Criteria:

* Past medical history of pacemaker implantation
* Pregnancy or lactating
* History of Atrial arrhythmia within the past year
* Elevated liver enzymes pre-operatively
* Past medical history of any liver disease or history of liver transplantation
* Use of statins or any anti-arrhythmics (including beta-blockers, calcium channel blockers, digoxin) within 3 months prior to surgery
* Pre-op EKG showing atrial arrhythmia

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Cerfolio, MD, Principal Investigator — University of Alabama at Birmingham, Department of Surgery
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 41 | 32
Completed | 30 | 25
Not Completed | 11 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Ineligible | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 41 | 32 | 73
Age Continuous [Median (Full Range); unit: years] | 62 [27 to 79] | 61 [30 to 81] | 61 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 41 | 32 | 73

OUTCOME MEASURES:

1. Primary Outcome: Atrial Fibrillation
Time Frame: 0-21 days post-operative
Measure: Number; unit: participants
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 30 | 25
participants | 6 | 1

ADVERSE EVENTS:
Arm/Group | Atorvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 11/30 | 3/25
Other Adverse Events (participants affected / at risk) | 25/30 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=30) | Placebo (N=25)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Subcutaneous Air (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Elevated Liver Function Tests (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Airleak (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=30) | Placebo (N=25)
Hypotension (Cardiac disorders) | 9 (9) | 1 (1)
Anemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 14 (14)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 25 (25) | 17 (17)
Airleak (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Tachycardia (Cardiac disorders) | 16 (16) | 11 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 22 (22) | 5 (5)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Indigestion (Gastrointestinal disorders) | 1 (1) | 3 (3)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Itching (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (12) | 6 (6)
Sub-Q Emphysema (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (7)
Atrial Fibrillation (Cardiac disorders) | 5 (5) | 1 (1)
Fever (General disorders) | 4 (4) | 3 (3)
Non-STEMI Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Elevated Troponin (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Insomnia (General disorders) | 3 (3) | 0 (0)
Tremors (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Lethargy (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes